CLINICAL TRIAL: NCT05079607
Title: A Modified Draize Repeat Insult Patch Test in a Shared Panel of 50/100 Healthy Volunteers, to Investigate the Irritation and Sensitization Potential of Test Articles Following Repeated Cutaneous Patch Applications
Brief Title: Human Skin Safety Testing of a Mitopure Topical Product Using a Human Repeat Insult Patch Test (HRIPT) in Healthy Volunteers
Acronym: GLOW-Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Princeton Research Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ASARIP1M
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Irritation/Irritant; Sensitisation
Keywords: HRIPT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitopure Topical Formula (Experimental)
  Interventions: Other: Mitopure Topical Formula 1; Other: Mitopure Topical Formula 2

INTERVENTIONS:
Other: Mitopure Topical Formula 1 — topical skin cream containing the low dose mitophagy activator Mitopure
Other: Mitopure Topical Formula 2 — topical skin cream containing the high dose mitophagy activator Mitopure

SUMMARY:
The objective of this study is to investigate the irritation and sensitization potential of multiple topically applied test articles (containing different concentrations of Mitopure), in a shared panel of healthy volunteers by means of repeated cutaneous patch applications under occlusion based on the modified Draize method

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females,18 years of age or older.
* Completed written informed consent.
* Female subject agrees to use an acceptable method of birth control (e.g. abstinence, condoms, hormonal birth control, IUD, tubal ligation, hysterectomy, bilateral oophorectomy, hysterectomy, post-menopausal for at least one year or male partner vasectomy).

Exclusion Criteria:

* Pregnancy or lactation.
* A current skin disease of any type apart from mild facial acne (e.g. eczema, psoriasis) or has tattoos or excessive hair at the patch sites that would interfere with patching/skin evaluations.
* Heavy alcohol consumption (i.e. more than 21 units per week or 8 units a day for men, more than 14 units per week or 4 units a day for women).
* Current use or history of repeated use of street drugs.
* A febrile illness lasting more than 24 hours in the six days prior to first patch application.
* Significant past medical history of hepatic, renal, cardiac, pulmonary, digestive, haematological, neurological, locomotor or psychiatric disease.
* Currently taking asthma medication or antihistamines for hay fever.
* A history of multiple drug hypersensitivity.
* Concurrent medication likely to affect the response to the test articles or confuse the results of the study (e.g. Anti-allergy, glucocorticoid, aspirin, non- steroidal anti-inflammatory, asthma or hay fever medication).
* Known sensitivity to the test articles or their constituents including patch materials (for example tape/plaster adhesive).
* Current treatment by a physician for allergy unless physician consulted by Investigator and participation approved.
* Participation in a repeat insult patch test (RIPT) or follow-up work within the last month.
* Sensitisation or questionable sensitisation in a RIPT.
* Recent immunisation (less than 10 days prior to test patch application).
* A medical history indicating atopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Skin safety as assessed by the number of adverse events of skin irritation and sensitization during human repeat insult patch testing (HRIPT) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, MD, PhD, Study Director — Amazentis SA
Locations (1):
- PCR Corp, 667A Stockport Road, Manchester, United Kingdom